CLINICAL TRIAL: NCT04536987
Title: Robot Therapy for Rehabilitation of Hand Movement After Stroke
Acronym: HEXORR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Catholic University of America (Other)
Collaborators: MedStar National Rehabilitation Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-315
Record Dates: First submitted 2020-07-29; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Movement Disorders; Hemiparesis
Keywords: robotic therapy; finger; hand
MeSH Terms: conditions — Stroke; Movement Disorders; Paresis

STUDY DESIGN:
Intervention Model Description: Random assignment to two study groups
Who Masked: Outcomes Assessor
Masking Description: Staff performing clinical evaluations was unaware of the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- low-dosage robot therapy (Experimental): 12 sessions of robotic therapy over 4-5 weeks
  Interventions: Device: HEXORR
- hi-dosage robot therapy (Experimental): 24 sessions of robotic therapy over 8-10 weeks
  Interventions: Device: HEXORR

INTERVENTIONS:
Device: HEXORR — The subject receives robotic assistance from the HEXORR robot during finger and thumb movements. Several different video games are used to provide feedback of performance and motivate the training. The assistance level is adjusted automatically in some games and manually in other games to enable a target success rate of 67% when playing the games.

SUMMARY:
A study will be performed where individuals with chronic stroke will be randomly assigned to receive 2 different dosages of robotic hand therapy. One group will receive 12 sessions of robot-assisted repetitive movement practice in the HEXORR robot over a 4-5 week period. A second group will receive 24 sessions of HEXORR therapy over a 8-10 week period.

DETAILED DESCRIPTION:
The overall goal of the proposed work is to improve hand function after stroke. Adequate hand function is critical to a functional upper limb, and is often resistant to conventional therapeutic interventions. Many stroke survivors have residual ability to flex the fingers, but extension is often limited and impeded by increased passive stiffness in flexors, involuntary activation of flexors and inability to activate extensors. The rationale for this approach stems from the growing evidence that neuro-rehabilitation after stroke may be enhanced via the application of motor learning strategies within the context of repetitive movement practice. The key therapeutic aspects of these strategies are high repetition, volitional effort, and successful completion of tasks to prevent frustration. While these represent promising therapeutic strategies, they are limited to mildly impaired subjects who already have enough control of finger extension to tolerate high repetitions of grasp/release tasks without succumbing to fatigue and/or frustration. There is a very large population of stroke patients who don't fall into this category and often must rely on compensatory strategies. In these patients, repetitive task practice facilitated by a robotic device may be more effective than unassisted task practice.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of stroke more than 6 months prior to randomization
2. presence of voluntary hand activity indicated by a score of at least 1 on the finger mass extension/grasp release item of the Fugl-Meyer Test of Motor Function
3. adequate cognitive status, as determined by Mini-Mental Status Examination score >24

Exclusion Criteria:

1. were under the influence of oral or injected antispasticity medications during the study
2. had MCP and IP passive extension limit > 30 degrees from full extension
3. had pain that interfered with daily activities
4. had excessive tone in the fingers and thumb as determined by Ashworth scores >=3
5. had severe sensory loss or hemispatial neglect as determined by clinical exam.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Test of Motor Function | 6 month follow-up
  Measures motor impairment in the upper extremity after stroke

SECONDARY OUTCOMES:
Change in Action Research Arm Test | 6 month follow-up
  Measures functional limitations of the upper extremity
Change in finger extension range of motion (degrees) | 6 month follow-up
  Motion capture of finger and thumb movement will be used to assess extension ability in units of degrees. The task will be to open the hand as far as possible from a closed fist. Data from all digits will be averaged to provide a single metric for extension ability of the fingers and thumb.
Change in Modified Ashworth Test | 6 month follow-up
  Measures hypertonia in the flexors of the fingers, wrist and elbow joints
Change in Motor Activity Log | 6 month follow-up
  Measures the amount of use of the upper extremity in ADL
Change in Grip Strength | 6 month follow-up
  Jamar Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lum, Principal Investigator — The Catholic University of America
Locations (1):
- MedStar National Rehabilitation Network, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data.

REFERENCES:
- [Background] Godfrey SB, Holley RJ, Lum PS. Evaluation of HEXORR Tone Assistance Mode Against Spring Assistance. IEEE Trans Neural Syst Rehabil Eng. 2015 Jul;23(4):610-7. doi: 10.1109/TNSRE.2015.2398933. Epub 2015 Feb 4. PMID 25667355
- [Background] Godfrey SB, Holley RJ, Lum PS. Clinical effects of using HEXORR (Hand Exoskeleton Rehabilitation Robot) for movement therapy in stroke rehabilitation. Am J Phys Med Rehabil. 2013 Nov;92(11):947-58. doi: 10.1097/PHM.0b013e31829e7a07. PMID 23900016
- [Background] Schabowsky CN, Godfrey SB, Holley RJ, Lum PS. Development and pilot testing of HEXORR: hand EXOskeleton rehabilitation robot. J Neuroeng Rehabil. 2010 Jul 28;7:36. doi: 10.1186/1743-0003-7-36. PMID 20667083